CLINICAL TRIAL: NCT04508075
Title: A Phase III, Observer-blind, Randomized, Placebo-controlled Study of the Efficacy, Safety and Immunogenicity of SARS-CoV-2 Inactivated Vaccine in Healthy Adults Aged 18-59 Years in Indonesia
Brief Title: Efficacy, Safety and Immunogenicity Study of SARS-CoV-2 Inactivated Vaccine
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Faculty of Medicine Universitas Padjadjaran (Unknown); National Intitute of Health Research and Development, Ministry of Health Republic of Indonesia (Unknown); Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CoV2-0320
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: SARS-CoV2 Infection
Keywords: vaccine; SARS-CoV-2; infection
MeSH Terms: conditions — COVID-19; Infections | interventions — COVID-19 Vaccines

STUDY DESIGN:
Intervention Model Description: Subjects 18-59 years of age: Randomized, observer blind, placebo-controlled two arms parallel group, prospective intervention study, to evaluate efficacy, safety, immunogenicity SARS-CoV-2 vaccine (inactivated)
Who Masked: Participant, Investigator
Masking Description: Observer blind Investigational Product and Active Comparator was masking Number of lot was masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SARS-CoV-2 Vaccine (Experimental): Participants receive 2 doses of SARS-CoV-2 Inactivated Vaccine with 14 days interval, intramuscularly
  Interventions: Biological: SARS-CoV-2 vaccine (inactivated)
- Placebo (Placebo Comparator): Participants receive 2 doses of placebo with 14 days interval, intramuscularly
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 vaccine (inactivated) — SARS-CoV-2 vaccine (inactivated) manufactured by Sinovac
  Arms: SARS-CoV-2 Vaccine
Biological: Placebo — Placebo manufactured by PT. Bio Farma
  Arms: Placebo

SUMMARY:
This phase III trial aims to assess the efficacy, safety and immunogenicity of SARS-CoV-2 Vaccine (inactivated) and lot-to-lot consistency evaluation

DETAILED DESCRIPTION:
This trial is Randomized, observer-blind, placebo-controlled two arms parallel group, prospective intervention study

Approximately 1620 subjects aged 18-59 years will be enrolled in this trial for efficacy evaluation. Subjects will be divided into 2 treatment arms that are the vaccinated group and placebo group with ratio 1:1. The vaccinated arms will be grouped into three different lot number (lot 1/lot 2/ lot 3) of SARS-CoV-2 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy adults aged 18 - 59 years.
2. Subjects have been informed properly regarding the study and signed the informed consent form.
3. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
2. Contact with novel coronavirus infected persons (positive for nucleic acid detection) within 14 days prior to the trial.
3. Contact to patients with fever or respiratory symptoms surrounding areas or from communities with reported cases within 14 days prior to the trial.
4. Two or more cases of fever and/or respiratory symptoms in a small area such as home, office, school and class within 14 days prior to the trial.
5. Evolving mild, moderate or severe illness, especially infectious disease or fever (body temperature ≥37.5℃, measured with infrared thermometer/thermal gun).
6. The result of RT-PCR of swab nasopharyngeal is positive
7. Reactive IgG and IgM for SARS-CoV-2 (by standardize rapid test).
8. Women who are lactating, pregnant or planning to become pregnant during the study period (judged by self-report of subjects and urine pregnancy test results).
9. History of asthma, history of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
10. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
11. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc) which according to the investigator might interfere with the assessment of the trial objectives.
12. Subjects who have any history of confirmed or suspected immunosuppressive or immunodeficient state, or received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long-term corticosteroid therapy (> 2 weeks)).
13. Subjects who have history of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain-Barre Syndrome
14. Subjects receive any vaccination within 1 month before and after IP immunization.
15. Subjects plan to move from the study area before the end of study period.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1620 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of laboratory-confirmed COVID-19 after the second dose | 14 days to 6 months after the second dose
  Percentage of laboratory-confirmed COVID-19 cases

SECONDARY OUTCOMES:
Incidence of suspected COVID-19 cases | within 14 days to 6 months after the second dose.
  Percentage of suspected COVID-19 cases
Incidence of laboratory-confirmed cases (severe, critical and death) | within 14 days to 6 months after the second dose
  Percentage of laboratory-confirmed cases (severe, critical, death)
Seroconversion rate anti-S antibody IgG titer (ELISA) | 14 days after two doses of vaccination
  Percentage of subjects with four-fold increasing anti-S antibody IgG titer (ELISA) compare to baseline and between batches
Seroconversion rate anti-S antibody IgG titer (ELISA) | 6 months after two doses of vaccination
  Percentage of subjects with four-fold increasing anti-S antibody IgG titer (ELISA) compare to baseline and between batches
Seropositive rate of neutralizing antibodies | 14 days after two doses of vaccination
  Percentage of subjects with four-fold increasing serum neutralizing antibody compared to baseline and between batches
Seropositive rate of neutralizing antibodies | 6 months after two doses of vaccination
  Percentage of subjects with four-fold increasing serum neutralizing antibody compared to baseline and between batches

OTHER OUTCOMES:
Local reaction and systemic events | 30 minutes to 14 days after each vaccination
  Number of Local reactions and systemic events
Local reaction and systemic events occurring after the last vaccination | 14 days to 28 days following last vaccination
  Number of Local reactions and systemic events
Serious adverse events during study | 6 months after the last dose
  Number of any SAE occur

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Sadikin Hospital/School of Medicine, Padjadjaran University, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Interim Result — https://doi.org/10.1016/j.vaccine.2021.09.052